CLINICAL TRIAL: NCT04219540
Title: Long-acting Buprenorphine vs. Naltrexone Opioid Treatments in CJS-involved Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-01450
Record Dates: First submitted 2019-11-26; First posted 2020-01-07 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- extended-release buprenorphine (XR-B) (Experimental): Subjects who agree to XR-B treatment will receive an XR-B injection to the abdomen. The injection is a liquid medication in the amount of either 100 or 300 mg buprenorphine in 1.5 cc volume and will last in the body for about 30 days. The medication is stored in a small nodule under the skin of the belly where it was injected. The buprenorphine is gradually released into the body over time for a 30-day period.
  Interventions: Drug: XR-B (SUBLOCADETM)
- extended release naltrexone XR-NTX (Experimental): Subjects who agree to XR-NTX treatment will receive an injection of XR-NTX to the outer upper part of your buttock. The injection is a liquid medication in the amount of 380 mg naltrexone in 4 cc volume (about 1 teaspoon) and will last in your body for about 30 days. Following release, visits with study physicians at Bellevue Hospital will offer further counseling or medication treatment referrals, the option to receive additional XR-NTX injections once a month following the first injection and continued encouragement to avoid relapses and stay on treatment.
  Interventions: Drug: XR-NTX
- Treatment as Usual (TAU) (No Intervention): In this group you will not receive any study medication. You will be able to receive any treatments available to individuals in the jail or prison who are not in the study. Trained study staff at the first two visits will provide counseling focusing on relapse and overdose prevention, treatment engagement, and navigating re-entry challenges.

INTERVENTIONS:
Drug: XR-B (SUBLOCADETM) — XR-B (SUBLOCADETM) contains buprenorphine, a partial opioid agonist, and is indicated for the treatment of moderate to severe opioid use disorder in patients who have initiated treatment with a transmucosal buprenorphine-containing product, followed by dose adjustment for a minimum of 7 days. Following induction and dose adjustment with sublingual buprenorphine, the recommended starting dose is 300 mg monthly for the first two months followed by a maintenance dose of 100 mg monthly thereafter. XR-B is administered monthly only by subcutaneous injection in the abdominal region. Study clinical staff will have flexibility to continue the 300mg dose for greater than 2 months, or use the 100mg dose for initial induction, if the participant's opioid use history or clinical status at the time of dosing support these decisions.
  Other Names: SUBLOCADE TM
  Arms: extended-release buprenorphine (XR-B)
Drug: XR-NTX — XR-NTX (Vivitrol®) produces a 30-day mu opioid receptor antagonist blockade Induction procedures require detoxification off opioids (5-7 days since last opioid use), a negative opioid urine toxicology, negative self-report of any recent opioid use, and a naloxone challenge. The naloxone challenge consists of 0.4-0.8mg of IV/SC/IM naloxone followed by the observation of no opioid withdrawal symptoms, or the use of oral naltrexone (12.5-25mg) followed by 1-2 hours of observation. XR-NTX is then delivered as a 380mg (4cc) intramuscular injection to the upper outer gluteus (buttock). Study interventions are FDA-approved, used in accordance with FDA-labeling and will be administered by a study clinician
  Other Names: Vivitrol®
  Arms: extended release naltrexone XR-NTX

SUMMARY:
This study seeks to compare the effectiveness of two medications used to treat opioid use disorder, extended-release buprenorphine (XR-B) vs. extended-release naltrexone (XR-NTX), among adults currently incarcerated in U.S. jails and prisons at 5 distinct trial sites. This open-label, non-inferiority, head-to-head study design will offer providers, correctional and public health authorities, payers and policy makers' timely and relevant data to assess the effectiveness of XR-B (and XR-NTX) as potentially useful re-entry and relapse prevention treatment options. It is hypothesized that XR-B is non-inferior to XR-NTX when comparing retention-in-study-medication treatment options.

DETAILED DESCRIPTION:
Participants eligible for randomization will be randomized 1:1 to extended-release buprenorphine (XR-B) vs. extended-release naltrexone (XR-NTX) prior to release from the correctional controlled environment (including jails, prisons, work release and residential treatment, or other correctional facilities) and treated for 24-weeks following release or upon entry into a community CJS-mandated program.

XR-B (SublocadeTM, Indivior) is a partial opioid agonist indicated for the treatment of moderate to severe opioid use disorder. Delivered as a pre-filled 2cc subcutaneous monthly injection, typically using two 300mg/1.5 ml initial starting doses followed by 100mg/0.5 ml monthly maintenance doses. The study will provide up to six monthly XR-B doses throughout the study. Prior to an initial injection, the participant must be stable for seven days or longer on sublingual buprenorphine (SLB) at doses of 8mg/day or higher.

Description of Study Intervention Participants eligible for randomization (n=670) will be randomized 1:1 to extended-release buprenorphine (XR-B) vs. extended-release naltrexone (XR-NTX) prior to release from the correctional controlled environment (including jails, prisons, work release and residential treatment, or other correctional facilities) and treated for 24-weeks following release or upon entry into a community CJS-mandated program.

XR-B (SublocadeTM, Indivior) is a partial opioid agonist indicated for the treatment of moderate to severe opioid use disorder. Delivered as a pre-filled 2cc subcutaneous monthly injection, typically using two 300mg/1.5 ml initial starting doses followed by 100mg/0.5 ml monthly maintenance doses. The study will provide up to six monthly XR-B doses throughout the study. Prior to an initial injection, the participant must be stable for seven days or longer on sublingual buprenorphine (SLB) at doses of 8mg/day or higher.

XR-NTX (Vivitrol®, Alkermes) is an opioid antagonist indicated for the prevention of opioid dependence, following detoxification. A negative opioid urine toxicology, negative self-report of any recent opioid use, and a naloxone challenge. The naloxone challenge consists of 0.4-0.8mg of IV/SC/IM naloxone followed by the observation of no opioid withdrawal symptoms, or the use of oral naltrexone (12.5-25mg) followed by 1-2 hours of observation. XR-NTX is delivered as a 380mg (4cc) intramuscular injection to the upper outer gluteus (buttock) monthly. The study will provide six or more monthly XR-NTX doses.

ELIGIBILITY:
Inclusion Criteria:

XR-B vs. XR-NTX Inclusions:

* (1) Adult volunteer aged 18 years or older able to provide written informed consent in English (or Spanish at some sites)
* (2) Current CJS incarceration (residing in a controlled environment) with pending release date (within 6 months of randomization) OR community CJS-involvement defined as: a) Current CJS incarceration (residing in a controlled environment) with pending release date (within 6 months of anticipated randomization), or; b) Community-dwelling volunteers with current CJS-involvement. [Current CJS-involvement is defined as either 1) release from any CJS incarceration or detention, or 2) under community supervision (includes parole, probation, drug or other treatment court, or other alternative to incarceration supervision) within 6 months prior to study enrollment (the date of a signed ICF)].
* (3) Current or history of moderate-to-severe opioid use disorder in the past year prior to incarceration (OUD, DSM-5)
* (4) Not planning to move out of state or to new location within 6-months post-release (reasonable chance they can complete 6 months of follow-up visits).
* (5) Willing to accept either XR-B or XR-NTX assignment.

Non-randomized TAU Inclusions:

• Recruited prior to launch of RCT or not interested in or appropriate for randomization to XR-B or XR-NTX assignment (i.e, already on methadone pre-release), but are otherwise eligible based on inclusion (#1-4, above) and exclusion (#6-10, below).

Exclusion Criteria:

XR-B vs. XR-NTX Exclusions:

* (6) Medical or psychiatric disorders making participation unsafe or regular follow-up unlikely, (such as suicidal ideation or pre-existing moderate to severe hepatic impairment)
* (7) Pregnancy, planning conception, or breast-feeding
* (8) Allergy, hypersensitivity or medical contraindication to either medication
* (9) Chronic pain requiring opioid pain management
* (10) On daily stable methadone or buprenorphine (SL-B) maintenance every day for past 30 days prior to incarceration or monthly XR-NTX or XR-BUP 30 days or longer prior to incarceration AND intending to remain on same form of methadone or buprenorphine or XR-NTX maintenance now and upon return to the community (i.e., was in MOUD treatment pre-incarceration, on same MOUD treatment now, and plans to continue same MOUD treatment post-incarceration). (Note - If community-dwelling, already on non-study methadone, buprenorphine, or naltrexone for 30 days or longer at the time of enrollment, and planning on continuing same.)

Non-randomized TAU Exclusions:

• Currently treated with non-study MOUD while currently incarcerated and for 30+ days prior to incarceration, or, if community-dwelling, currently on MOUD for 30 days or longer at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Number of Injections during 24-Week Post-Release Treatment Phase | Up to Week 24
  The primary outcome measure is retention-in-study-medication-treatment post-release during weeks 1-24; retention is defined as the proportion of scheduled study medication injections received. The total score ranges from 0-6 and is scored as following: less than 6 XR-B injections will contribute to lower retention (<5 of 6), and 7+ XR-NTX will contribute only to maximum retention (6 of 6).

SECONDARY OUTCOMES:
Change in Opioid use | Weeks 0, 4, 8, 12,16, 20, 24, 52
  Change in opioid treatment outcomes will assess for illicit opioid use through self-reported opioid use (days per month), opioid-positive urine samples (negative vs. positive or missing, monthly), and overdose events (fatal and non-fatal),
Change in Opioid treatment outcomes - adverse events | Weeks 0, 4, 8, 12,16, 20, 24, 52
  Change in Opioid use will be tracked monthly through non-fatal and fatal overdose events and other adverse events and death recorded on the Opioid Overdose AE form and the Opioid relapse outcome form.
Change in Opioid treatment outcomes - lifestyle changes | Weeks 0, 4, 8, 12,16, 20, 24, 52
  Non-study addiction treatment participation, depression scores (Hamilton Depression scale) and quality of life (WHOQOL) changes will be assessed for demographic, housing, employment status changes.
Change in Opioid treatment outcomes - HIV changes | Weeks 0, 24
  Changes in HIV sex and IVDU risk scores as well as HIV and HCV status will be assessed HIV/HCV risk behaviors (RAB), HIV P24ag/ ab with reflex HIV RNA (if HIV ab negative at baseline; if HIV AB positive at baseline just check HIV RNA) and HCVAb with reflex HCV RNA if AB positive ( if AB + at baseline then just HCV VL at f/u timepoints) at baseline week 24 and week 52
Change in criminal justice system (CJS) involvement with XR-B versus XR-NTX | Weeks 4, 8, 12,16, 20, 24, 52
  Criminal justice system (CJS) involvement and recidivism outcomes will be measured by the number of new criminal charges, new arrests, re-incarceration episodes, and re-incarceration days by CJS public records audits. XR-B may be an effective CJS intervention alongside other OUD medications and may ultimately allow for much wider uptake of opioid agonist medication treatments in CJS populations in comparison to XR-NTX.
Change in Non-randomized Treatment-As-Usual retention compared to XR-B/XR-N. | Weeks 4, 8, 12,16, 20, 24, 52
  TAU participants in this trial will be followed similarly to randomized participants but will not receive study medication or active medical treatment from the study. Prior to release from correctional controlled environment and at research visit follow-up in the community, all TAU participants will be provided education and materials that include information on opioid overdose prevention and referrals to other community addiction treatment services. TAU participants will receive the same visit incentives and study team contact, including Tracker services, as randomized participants. This amount of contact, incentives, education, and referrals are likely in excess than actual real-world 'usual care' of opioid use disorder patients released from a CJS controlled environment, and is in keeping with ethical standards for clinical trials among prisoners, in which all experimental arms must receive some tangible yet non-coercive benefit beyond usual care.
Change in Non-randomized Treatment-As-Usual rates of OUD | Weeks 4, 8, 12,16, 20, 24, 52
  TAU participants, particularly those not in treatment with an OUD medication, may well face higher risk of relapse and overdose vs. active randomized participants receiving study medications. TAU participants, particularly those not in treatment with an OUD medication, may well face higher risk of relapse and overdose vs. active randomized participants receiving study medications.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Lee, MD, Principal Investigator — NYU Langone
Locations (6):
- United States (6):
  - Yale University School of Medicine, New Haven, Connecticut
  - Friends Research Institute, Baltimore, Maryland
  - Dartmouth College, Hanover, New Hampshire
  - Rutgers University, New Brunswick, New Jersey
  - NYU Langone Health, New York, New York
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Upon reasonable request. Requests should be directed to mia.malone@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT04219540/ICF_000.pdf